CLINICAL TRIAL: NCT04121325
Title: Gastric Electrical Stimulation for Treating Abdominal Pain in Patients With Gastroparesis
Brief Title: Gastric Electrical Stimulation for Abdominal Pain in Gastroparesis
Status: Terminated | Type: Observational
Why Stopped: pandemic
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Thomas Abell, Professor, University of Louisville
Other Study IDs: 19.0915
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Gastroparesis patients with abdominal pain: Patients with gastroparesis who have had an Enterra device in place for at least two months who continue to have moderate to severe abdominal pain.
  Interventions: Device: Enterra

INTERVENTIONS:
Device: Enterra — To measure validated and subjective pain scores among patients with an existing GES device, and who have a trial of new settings directed at abdominal pain and compare their pain scores to each patient baseline symptoms, done with their previous GES settings.

SUMMARY:
To conduct a pilot study to evaluate the effects of new GES programming settings on abdominal pain in patients with gastroparesis and existing GES devices, whose abdominal pain has so far been refractory to drugs and/or devices.

DETAILED DESCRIPTION:
Eligible patients will undergo detailed pain assessments as well as non-invasive physiologic assessment. Patients existing GES devices will be reprogrammed to new setting for 4 week and their GI symptoms including pain will be evaluated by a daily diary. At the end of 4 weeks detailed pain assessments and noninvasive physiologic assessments will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Should be able to give informed consent for the study
* Has Enterra GES device in place for at least 2 months
* Continue to have moderate to severe abdominal pain on at least one pain questionnaire or >5 score (on a scale of 0-10 for pain) on the VAS questionnaire for at least 2 months.
* Abdominal pain should be either persistent; for example, daily for at least >1 hour, be chronic for >2 months, and refractory to original Enterra GES settings

Exclusion Criteria:

* Unable to provide informed consent
* Pregnancy
* Any other active health problems that would render patient unable to complete the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastroparesis patients with abdominal pain.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain | 4 weeks
  Abdominal Pain by Brief Pain Inventory. The values are 0-10, with 10 being worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Abell, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States